CLINICAL TRIAL: NCT02659852
Title: A Prospective Randomized Study for Efficacy of Side-by-side Compared to Stent-in-stent Technique in the Endoscopic Management of Malignant Hilar Biliary Obstruction
Brief Title: A Study for Efficacy of Side-by-side Compared to Stent-in-stent Technique in the Endoscopic Management of Malignant Hilar Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-1072
Record Dates: First submitted 2016-01-12; First posted 2016-01-20 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Cholangiocarcinoma; Gallbladder Cancer; Pancreatic Cancer; HCC; AOV Cancer
Keywords: Hilar malignant biliary obstruction; bilateral metal stent; stent in stent; side by side
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Pancreatic Neoplasms | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Side by side group (Experimental)
  Interventions: Procedure: side by side
- Stent in stent group (Active Comparator)
  Interventions: Procedure: stent in stent

INTERVENTIONS:
Procedure: side by side — Stenting generally begins with selective guidewire cannulation into the left and right intrahepatic bile ducts. Self-expandable metallic stent(SEMS) deployment is the conventional method and parallel SEMS can be inserted. SEMS deployment can be performed serially or simultaneously.
  Arms: Side by side group
Procedure: stent in stent — After first SEMS deployment, contralateral placement of a second SEMS through the mesh of the first deployed stent was done and it looks like a Y configuration.
  Arms: Stent in stent group

SUMMARY:
Malignant obstructive jaundice is a common complication of advanced stage cholangiocarcinoma, GB cancer, and pancreatic cancer. In biliary stricture by malignancy, biliary drainage with placement of self-expanding metal stent (SEMS) for palliation is the therapy of choice in these patients. On hilar biliary malignant obstruction, bilateral stent used to be inserted. There are two kinds of bilateral metal stent insertion methods in hilar biliary malignant obstruction. (Stent in stent vs. side by side) Previously, two studies was conducted to show the superiority of bilateral metal stent insertion between stent in stent and side by side. Biliary drainage and stent patency was a little superior in side by side than stent in stent. But, complication related with bilateral metal stent was increased in patients with side by side method. Another study showed that there was no significant difference between those bilateral stent insertion methods. The most important concern about side by side method is associated with portal vein thrombosis by bilateral stent diameter. Selection of proper stent insertion method in patients with hilar malignant biliary obstruction is still controversial.

The purpose of this study is to investigate the patency of stent and survival of patients in side by side method (6mm sized M type) compared to stent in stent method (10mm sized LCD type) in patient with hilar malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed hilar malignant biliary obstruction or clinically defined malignant biliary obstruction
* older than 20 years old

Exclusion Criteria:

* Operable case
* Non-hilar biliary malignant obstruction
* Duodenal obstruction
* Other cancer except biliary malignancy
* uncontrolled infection status
* Eastern Cooperative Oncology Group ≥ 3
* No signed informed consent
* Failed endoscopic approach to duodenum or biliary tract

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Median patency duration | 1 year after stent insertion
  Median patency duration from stent insertion date to stent occlusion date or last follow up date if stent is patent

SECONDARY OUTCOMES:
Overall survival | 1 year
complication rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Law R, Baron TH. Bilateral metal stents for hilar biliary obstruction using a 6Fr delivery system: outcomes following bilateral and side-by-side stent deployment. Dig Dis Sci. 2013 Sep;58(9):2667-72. doi: 10.1007/s10620-013-2671-4. Epub 2013 Apr 27. PMID 23625287
- [Background] Kim KM, Lee KH, Chung YH, Shin JU, Lee JK, Lee KT, Shim SG. A comparison of bilateral stenting methods for malignant hilar biliary obstruction. Hepatogastroenterology. 2012 Mar-Apr;59(114):341-6. doi: 10.5754/hge11533. PMID 22353496